CLINICAL TRIAL: NCT06453785
Title: Comparing pOrtable MRI and TRUS-Fusion Prostate Biopsy to Assess aCcuracy of Prostate Cancer Detection
Acronym: IP10-COMPACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22CX7739
Record Dates: First submitted 2024-04-25; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
Keywords: biopsy; MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients with suspected prostate cancer (Other): Patients who undergo prostate biopsy for suspected prostate cancer. Each patient would undergo both a portable MRI-registered biopsy and a TRUS-image-fusion biopsy. To reduce the risk of bias between the two modalities, the order of the modality will be randomized 1:1. There will be no blinding of the surgeon.
  Interventions: Device: Promaxo portable MRI

INTERVENTIONS:
Device: Promaxo portable MRI — The Promaxo portable MRI is an FDA cleared MRI device for MR-guided procedures. It uses a novel "truly" open MRI with an unobstructed field of view and central aperture for robotic guided intervention and has a limited footprint allowing it to be places in a standard operating theatre or large clinic room. The strength of magnet is also low enough that special precautions and equipment are not to take biopsies.

SUMMARY:
Currently, patients suspected of having prostate cancer undergo an MRI followed by targeted biopsies of any suspicious lesions under trans-rectal ultrasound (TRUS) guidance. This pathway is labour, time, and cost-intensive. Additionally, TRUS-MRI-Fusion devices are needed, which overlay the MRI scan onto the TRUS used for biopsies. This can lead to targeting errors due to mismatched images. Although biopsies can be performed in the MRI scanner to reduce these errors, it requires a significant amount of time within an expensive MRI scanner in the radiology department, along with special MRI-compatible equipment. Portable MRI technology has the potential to reduce these errors and streamline the diagnostic pathway to one visit. The Promaxo portable MRI is an FDA-cleared MRI device for MR-guided procedures. It uses a novel "truly" open MRI with an unobstructed field of view and a central aperture for robotic-guided intervention and has a limited footprint, allowing it to be placed in a standard operating theatre or large clinic room. The strength of the magnet is also low enough that special precautions and equipment are not needed to take biopsies.

The intention is to conduct a study that answers the following research question: How does the accuracy of targeted biopsies of the prostate performed under the guidance of a portable MRI scanner compare to TRUS-MRI-fusion biopsies?

Design: A single-arm, single-center IDEAL stage 2a study (n=85 patients) of patients undergoing prostate biopsy for suspected prostate cancer, where each patient would undergo both a portable MRI-registered biopsy and a TRUS-image-fusion biopsy. To reduce the risk of bias between the two modalities, the order of the modality will be randomized 1:1. There will be no blinding of the surgeon.

The primary outcome will be the technical feasibility of performing portable MRI and portable MRI-targeted biopsies and estimates on cancer detection.

DETAILED DESCRIPTION:
Design: A single arm, singe centre study of 85 patients who have been selected to undergo prostate biopsy for suspected prostate cancer. Each patient would undergo both a portable MRI registered biopsy and the local standard ultrasound fusion biopsy. To reduce the risk of bias between the two types of biopsy the sequence will be randomised 1:1. There will be no blinding of the surgeon.

Patient Journey:

Patients eligible for the study will have already undergone a standard of care prostate MRI and offered a biopsy for any suspicious lesions seen. Eligible Patients will initially be contacted by a member of the study team and given written information on the study, After a period of time for the patient to review the information the patient will be contacted to give consent which can either be performed remotely or face-to-face.

After consent they will be asked to fill in questionnaires for baseline genito-urinary and bowel function using validated questionnaires and overall health status; this will be online or via paper copies. The questionnaires will consist of the HADS score questionnaire, EPIC (urinary, erectile, bowel) questionnaires and EuroQoL [EQ-5D-5L].

Patients who have consented to the study will then undergo a combined biopsy procedure either under local anaesthetic or if the patient wishes under sedation or general anaesthetic.

The current biopsy standard operating procedure (SOP) requires that 6 targeted cores per-lesion are taken along with 10-12 systematic cores of the remaining prostate. To ensure patient do not have cores taken in excess of the local SOP each enrolled patient will undergo transperineal prostate biopsy under local anaesthetic or sedation/general anaesthetic with a total of 6-targeted cores taken per lesion (three using each biopsy modality, ultrasound fusion or Portable MRI). All suspicious lesions will biopsied.

The patient will then be seen again in either in clinic (remote or face to face) to be given their biopsy results 2-12 weeks after the biopsy. The time point for this appointment will depend on the processing time of the biopsies by the pathology department as per the local standard of care clinical pathway. At this visit patients will be asked again to fill in questionnaires for baseline genito-urinary and bowel function using validated questionnaires and overall health status; this will be online or via paper copies. The questionnaires will consist of the HADS score questionnaire, EPIC (urinary, erectile, bowel) questionnaires and EuroQoL [EQ-5D-5L]. All the above visits mirror the local standard of care clinical pathway and except for the consent visit which could take place on the same day of the biopsy if the patient wishes there will be no additional burden of visits upon the patient.

There will be some optional consent points:

First, patients will also be asked to give optional consent for identifiable data to be linked with the national databases (ONS and HES database). Subsequent funding will be applied for from academic and charity funders to allow to carry out the linkage work. The identifiable fields (NHS number) required for linkage will be encrypted using a one-way encryption algorithm. Patients will be asked if they are happy to give consent for their health status to be followed up over time. This will be done by linking their name and NHS number with records held by the NHS and maintained by the NHS Information Centre and NHS Central Register or any applicable NHS information system.

This will allow to track what happens after the study finishes and observe if anyone gets cancer in future and about the type of cancer and treatment they have had. Patients will be asked whether or not they give permission to be contacted by member of the study research team within 10 years of signing their health status (including details of any other tests and treatment they have had since the study) and quality of life. If the patient decides to take part a member of the study research team may send this request to the patient's home address. The intention is to link individual trial informationto national databases on cancer diagnosis, GP databases on healthcare and medication use and finally death registry to see if any of the men died from prostate cancer.

As prostate cancer is often a slow-growing disease which may not progress for many years, patients will also be asked if they are happy to keep personal data stored or accessed for 10 years on the NHSCR (National Health Service Care Register). Second, in order to get an area based estimate of deprivation, the participants' partial postcodes will be converted into an Index of Multiple Deprivation (IMD) score. The IMD is the established index of deprivation for England and Wales and has been adopted widely in studies across local and national government. Partial postcodes will be stored in the study database, only IMD rank, which is based on detailed ward-level index of deprivation based on severe separate domains.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above (no upper limit)
* Raised age specific PSA
* LIKERT/PIRADS 3 or above lesion on prostate mpMRI who have been advised to undergo a prostate biopsy.

Exclusion Criteria:

* Patients who are unable to undergo a diagnostic standard of care MRI due to metallic implants, foreign body or devices.
* Patients with a Cardiac pacemaker or Implantable cardioverter-defibrillator (ICD).
* Contraindication to performing a biopsy guided by a transrectal ultrasound probe
* Unable to give informed consent to the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Clinicical Significance of Cancer Detected | 2 years
  The proportion of patients with biopsy cores that yield cancer-positive results and the concordance between MRI-guided biopsy results and histopathological findings.
Technical feasibility of performing portable MRI and portable MRI targeted biopsies. | 2 years
  Percentage of biopsy completed

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 is a standardized system for grading the severity of adverse events (AEs) in clinical trials and medical practice. In CTCAE v4.0, adverse events are graded on a scale from Grade 1 to Grade 5, with each grade indicating increasing severity:
  Grade 1: Mild AE Grade 2: Moderate AE Grade 3: Severe or medically significant but not immediately life-threatening AE Grade 4: Life-threatening consequences AE Grade 5: Death related to AE
Patient reported outcome measures (PROMS / HADS-D) of genitourinary health | 2 years
  Hospital Anxiety and Depression Scale (HADS): Consists of 14 items, seven for anxiety (HADS-A) and seven for depression (HADS-D), scored on a Likert scale from 0 to 3. Higher scores indicate more anxiety or depression. Clinically significant levels are defined by cutoff scores.
Overall health-related quality of life as assessed by ICIQ-UI short form | 2 years
  The International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI SF) is a validated questionnaire used to assess the impact of urinary incontinence on an individual's health-related quality of life (HRQoL). It specifically focuses on the experience of urinary incontinence, including its frequency, severity, and the degree to which it affects daily activities and emotional well-being.
  The total score can be used to classify the severity of urinary incontinence:
  0-5: Slight or no impact 6-12: Moderate impact 13-18: Severe impact 19-21: Very severe impact
Overall health-related quality of life as assessed by IPSS | 2 years
  The International Prostate Symptom Score (IPSS) provides a quantitative measure of urinary symptoms, helping clinicians evaluate symptom severity and monitor changes over time.ach question in the IPSS is scored on a Likert scale from 0 to 5, with higher scores indicating greater symptom severity. The total IPSS score is calculated by summing the scores for the individual questions, resulting in a total score ranging from 0 to 35.
  Mild: 0-7 Moderate: 8-19 Severe: 20-35
Overall health-related quality of life as assessed by IPSS-QoL | 2 years
  International Prostate Symptom Score-Quality of Life assesses the impact of lower urinary tract symptoms (LUTS) on a patient's quality of life (QoL) specifically related to urinary symptoms associated with benign prostatic hyperplasia (BPH) or prostate enlargement. The IPSS-QoL consists of a single question that asks the patient to rate their perception of how urinary symptoms have affected their quality of life during the past month. The question is scored on a Likert scale from 0 to 6, with the following response options:
  Delighted (scored as 0) Pleased (scored as 1) Mostly satisfied (scored as 2) Mixed (about equally satisfied and dissatisfied) (scored as 3) Mostly dissatisfied (scored as 4) Unhappy (scored as 5) Terrible (scored as 6)
Overall health-related quality of life as assessed by EQ5D | 2 years
  EuroQol 5-Dimension (EQ-5D) assesses overall health status. Its questionnaire has two components: Descriptive System evaluates health across five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, and Anxiety/depression, each with three severity levels. This yields 243 possible health states. Visual Analog Scale (VAS) rates overall health from 0 (worst imaginable) to 100 (best imaginable).
The sensitivity, specificity, and accuracy of using portable MRI to detect clinically significant prostate cancer | 2 years
  Detection of clinically significant prostate cancer defined as Gleason grade 3+4 or greater and/or a maximum cancer core length of >/= 4mm.
  Detection of clinically significant prostate cancer defined as Gleason grade 4+3 or greater and/or a maximum cancer core length of >/= 6mm.
  This outcome will measure the sensitivity, specificity, and accuracy of portable MRI in detecting prostate cancer deemed clinically significant. Sensitivity refers to the proportion of true positive cases detected by the portable MRI, while specificity refers to the proportion of true negative cases correctly identified as negative. Accuracy measures the overall correctness of the portable MRI's detection compared to a standard MRI, or histopathology from biopsy samples.
Concordance Rate of Prostate Cancer Detection between Portable MRI and Standard mpMRI | 2 years
  A matched cohort of mpMRI, portable MRI, targeted and systematic biopsies will be created to estimate concordance of portable MRI compared to mpMRI in the detection of clinically significant cancer. Data from this analysis will allow the development of much larger RCT and screening study.
Patient reported outcome measures (PROMS / EPIC) of genitourinary health | 2 years
  EPIC (urinary, erectile, bowel): Expanded Prostate Cancer Index Composite. The score range is usually from 0 to 100. Higher scores denote better function and quality of life in respective domains.
Patient reported outcome measures (PROMS / EuroQol) of genitourinary health | 2 years
  EuroQol (EQ-5D-5L): EuroQol 5-Dimension 5-Level Scale. Assessing mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Responses range from no problems to extreme problems. VAS ranges from 0 to 100, reflecting worst to best imaginable health.

CONTACTS AND LOCATIONS:
Overall Officials: Taimur Shah, Dr, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No